CLINICAL TRIAL: NCT05659706
Title: Effectiveness of the Jeanne et Léon Program® on the Residents's Frailty in Temporary
Acronym: FRAQOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jeanne et Leon Developpement (Other)
Collaborators: Gerontopôle des Pays de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 21-S01
Record Dates: First submitted 2022-11-28; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Residents's Frailty in Temporary Accommodation; Residents's Quality of Life in Temporary Accommodation
Keywords: Frailty; Quality of life; Health event
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: "intervention" group, named "Group 3+": attend at least three workshops per week
  Interventions: Other: cognitive evaluations and non cognitive evaluations
- Arm 2: "control" group, named "Group 0-1": not participate in the activities program or will attend a maximum of one workshop per week.
  Interventions: Other: cognitive evaluations and non cognitive evaluations

INTERVENTIONS:
Other: cognitive evaluations and non cognitive evaluations — Mini Mental State Examination Charlson Comorbidity Index Katz Index ICOPE step 1 The 15-item geriatric depression scale (GDS-15) Medical Outcomes Study Short Form 36 (SF-36) Short Physical Performance Battery ( SPPB)

SUMMARY:
The management of frailty is a difficulty in the Temporary Accommodation Residences. Frailty represents a risk of reducing the activities of the elderly person. Jeanne & Léon Développement® offers an activity program that integrates several dimensions (physical and/or nutritional and/or social and/or psychological). To obtain the expected benefit, effect of the Jeanne & Léon® activities program on the residents's frailty and quality of life in temporary accommodation, the activity of at least one of these approaches is used as a global stimulant and thus activates the remaining skills to help fight against the frailty syndrome. In order to do this, the framework of the temporary accommodation, the group dynamics and the presence of a professional facilitator ensure the conditions for adherence to the program and promote the realization of stimulating activities.

The phenomenon of activation initiated during the residential activity program can lead to an improvement in the components of frailty which is maintained over time. This will be assessed in terms of the occurrence of events after the activity program has been followed.

DETAILED DESCRIPTION:
The clinical assessment will be performed by the investigating physician.

Initial follow-up: Fragility and Quality of Life assessment is carried out by the trained nursing staff (doctor, nurse) of the Résidence Les Tamaris. The clinical assessment will include screening for thymic disorders. All experimenters will be specifically trained in the protocol and GCP beforehand.

V0 (inclusion visit carried out within 72 hours after admission to the residence): inclusion after information and non-opposition, then randomization into the control group or the intervention group V1 (initial assessment visit performed within 96 hours after admission to the residence): initial assessment of the resident V2 (V1+ 21 days +/- 1 day: end of main study visit): final evaluation of the main study.

In case of discharge from the Residence: validation of the contact information and the follow-up telephone schedule of the participant.

Post-program follow-up: identification of intercurrent events by the Residence staff

VS1 (V2 + 1 Month), SV2 (V2 + 3 Months): interview of participants by on-site follow-up or telephone call VS3 (V2 + 6 Months): on-site follow-up or final phone call.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years and over
* Participant who has been living in temporary accommodation at the Résidence Les Tamaris for a maximum of 72 hours
* Visual, auditory and oral or written abilities in French sufficient to complete the assessments and participate in the Jeanne & Léon® Program activities
* Agrees to participate in the study and follow-ups for up to six months after the end of the activity program/temporary residence
* Non-opposition accompanied by the information note co-signed by the investigator and the resident participating in the study, or the family member or the designated trusted person (if applicable)
* Must be affiliated to a social security plan

Exclusion Criteria:

* Refusal to participate by the resident, family member or designated support person
* Communication difficulties, sensory and/or motor deficits
* Medical contraindication
* Participant already included in another research protocol
* Person under legal protection

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will focus on elderly people (men and women) living in temporary accommodation in the Résidence Les Tamaris.
  It will take place in the residents' living quarters.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
The endpoint will be a composite score, the FRAQOL, based on a combination of functional performance assessment (Short Physical Performance Battery (SPPB) composite test) and Quality of Life (Short Form 36 (SF-36) self questionnaire). | 8 months
  The endpoint will be a composite score, the FRAQOL, based on a combination of functional performance assessment (Short Physical Performance Battery (SPPB) composite test) and Quality of Life (Short Form 36 (SF-36) self questionnaire).
  The Short Physical Performance Battery (SPPB) composite test and Short Form 36 (SF-36) self questionnaire will be assessed within 96 hours of admission to the residence, prior to program implementation, and then 3 weeks after the initial assessment
  SPPB: minimum value = 0 ; maximum value = 12 SPPB 0-6= Low performance SPPB 7-9 =Intermediate intermédiaires SPPB 10-12 =High performance
  SF36: minimum value = 0 ; maximum value = 100

SECONDARY OUTCOMES:
Evolution of each item of the scores Short Form 36 self questionnaire | 15 months
  Evolution of each item of the scores Short Form 36 self questionnaire
Evolution of each item of the scores Short Physical Performance Battery (SPPB) composite test | 15 months
  Evolution of each item of the scores Short Physical Performance Battery (SPPB) composite test
Evolution of each item of the Step 1 of ICOPE(Integrated Care for Older People) | 15 months
  Evolution of each item of the Step 1 of ICOPE(Integrated Care for Older People)
  no scores: answers yes/no to different items
Evolution of intercurrent health events of the composite score FRAQOL at one, three and six months after the end of the program | 15 months
  Evolution of intercurrent health events of the composite score FRAQOL at one, three and six months after the end of the program The objective is to estimate the frequency of occurrence of intercurrent health events of the composite score FRAQOL
Estimation of the incremental cost associated with the occurrence of intercurrent events up to six months after program completion | 15 months
  Estimation of the incremental cost associated with the occurrence of intercurrent events up to six months after program completion
Use of the ICOPE screening questionnaire responses as a descriptive element of the study population and analysis of a potential predictive relationship on the 6-month outcome. | 15 months
  Use of the ICOPE screening questionnaire responses as a descriptive element of the study population and analysis of a potential predictive relationship on the 6-month outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BERRUT, Pr, Study Director — Gérontopôle des Pays de la Loire
Locations (1):
- Résidence les Tamaris- Jeanne et Léon Développement, Bois-de-Céné, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tinetti ME, Fried T. The end of the disease era. Am J Med. 2004 Feb 1;116(3):179-85. doi: 10.1016/j.amjmed.2003.09.031. PMID 14749162
- [Background] Rolland Y, Benetos A, Gentric A, Ankri J, Blanchard F, Bonnefoy M, de Decker L, Ferry M, Gonthier R, Hanon O, Jeandel C, Nourhashemi F, Perret-Guillaume C, Retornaz F, Bouvier H, Ruault G, Berrut G. [Frailty in older population: a brief position paper from the French society of geriatrics and gerontology]. Geriatr Psychol Neuropsychiatr Vieil. 2011 Dec;9(4):387-90. doi: 10.1684/pnv.2011.0311. French. PMID 22182814
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] The World Health Organization Quality of Life Assessment (WHOQOL): development and general psychometric properties. Soc Sci Med. 1998 Jun;46(12):1569-85. doi: 10.1016/s0277-9536(98)00009-4. PMID 9672396
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Hunt SM, McKenna SP, McEwen J, Williams J, Papp E. The Nottingham Health Profile: subjective health status and medical consultations. Soc Sci Med A. 1981 May;15(3 Pt 1):221-9. doi: 10.1016/0271-7123(81)90005-5. No abstract available. PMID 6973203
- [Background] Vagetti GC, Barbosa Filho VC, Moreira NB, Oliveira Vd, Mazzardo O, Campos Wd. Association between physical activity and quality of life in the elderly: a systematic review, 2000-2012. Braz J Psychiatry. 2014 Jan-Mar;36(1):76-88. doi: 10.1590/1516-4446-2012-0895. Epub 2014 Jan 17. PMID 24554274
- [Background] Perneger TV, Leplege A, Etter JF, Rougemont A. Validation of a French-language version of the MOS 36-Item Short Form Health Survey (SF-36) in young healthy adults. J Clin Epidemiol. 1995 Aug;48(8):1051-60. doi: 10.1016/0895-4356(94)00227-h. PMID 7775992
- [Background] Leplege A, Ecosse E, Verdier A, Perneger TV. The French SF-36 Health Survey: translation, cultural adaptation and preliminary psychometric evaluation. J Clin Epidemiol. 1998 Nov;51(11):1013-23. doi: 10.1016/s0895-4356(98)00093-6. PMID 9817119
- [Background] de Lira CAB, Taveira HV, Rufo-Tavares W, Amorim ADS, Ferreira LMC, Andrade MS, Vancini RL. Engagement in a Community Physical Activity Program and Its Effects Upon the Health-Related Quality of Life of Elderly People: A Cross-Sectional Study. Value Health Reg Issues. 2018 Dec;17:183-188. doi: 10.1016/j.vhri.2018.10.002. Epub 2018 Nov 9. PMID 30419539
- [Background] Rosenberg T, Montgomery P, Hay V, Lattimer R. Using frailty and quality of life measures in clinical care of the elderly in Canada to predict death, nursing home transfer and hospitalisation - the frailty and ageing cohort study. BMJ Open. 2019 Nov 12;9(11):e032712. doi: 10.1136/bmjopen-2019-032712. PMID 31722953
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310
- [Background] Marzetti E, Calvani R, Tosato M, Cesari M, Di Bari M, Cherubini A, Broccatelli M, Savera G, D'Elia M, Pahor M, Bernabei R, Landi F; SPRINTT Consortium. Physical activity and exercise as countermeasures to physical frailty and sarcopenia. Aging Clin Exp Res. 2017 Feb;29(1):35-42. doi: 10.1007/s40520-016-0705-4. Epub 2017 Feb 8. PMID 28181204
- [Background] Landi F, Abbatecola AM, Provinciali M, Corsonello A, Bustacchini S, Manigrasso L, Cherubini A, Bernabei R, Lattanzio F. Moving against frailty: does physical activity matter? Biogerontology. 2010 Oct;11(5):537-45. doi: 10.1007/s10522-010-9296-1. Epub 2010 Aug 10. PMID 20697813
- [Background] Bauman A, Merom D, Bull FC, Buchner DM, Fiatarone Singh MA. Updating the Evidence for Physical Activity: Summative Reviews of the Epidemiological Evidence, Prevalence, and Interventions to Promote "Active Aging". Gerontologist. 2016 Apr;56 Suppl 2:S268-80. doi: 10.1093/geront/gnw031. PMID 26994266
- [Background] Teri L, Gibbons LE, McCurry SM, Logsdon RG, Buchner DM, Barlow WE, Kukull WA, LaCroix AZ, McCormick W, Larson EB. Exercise plus behavioral management in patients with Alzheimer disease: a randomized controlled trial. JAMA. 2003 Oct 15;290(15):2015-22. doi: 10.1001/jama.290.15.2015. PMID 14559955
- [Background] Geirsdottir OG, Arnarson A, Briem K, Ramel A, Tomasson K, Jonsson PV, Thorsdottir I. Physical function predicts improvement in quality of life in elderly Icelanders after 12 weeks of resistance exercise. J Nutr Health Aging. 2012 Jan;16(1):62-6. doi: 10.1007/s12603-011-0076-7. PMID 22238003
- [Background] Park SY, Kim JK, Lee SA. The effects of a community-centered muscle strengthening exercise program using an elastic band on the physical abilities and quality of life of the rural elderly. J Phys Ther Sci. 2015 Jul;27(7):2061-3. doi: 10.1589/jpts.27.2061. Epub 2015 Jul 22. PMID 26311926
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Cho KO. The Positive Effect of Physical Activity on Health and Health-related Quality of Life in Elderly Korean People-Evidence from the Fifth Korea National Health and Nutrition Examination Survey. J Lifestyle Med. 2014 Sep;4(2):86-94. doi: 10.15280/jlm.2014.4.2.86. Epub 2014 Sep 30. PMID 26064859
- [Background] Aoki K, Sakuma M, Ogisho N, Nakamura K, Chosa E, Endo N. The effects of self-directed home exercise with serial telephone contacts on physical functions and quality of life in elderly people at high risk of locomotor dysfunction. Acta Med Okayama. 2015;69(4):245-53. doi: 10.18926/AMO/53561. PMID 26289916
- [Background] Liposcki DB, da Silva Nagata IF, Silvano GA, Zanella K, Schneider RH. Influence of a Pilates exercise program on the quality of life of sedentary elderly people: A randomized clinical trial. J Bodyw Mov Ther. 2019 Apr;23(2):390-393. doi: 10.1016/j.jbmt.2018.02.007. Epub 2018 Feb 11. PMID 31103125
- [Background] Lok N, Lok S, Canbaz M. The effect of physical activity on depressive symptoms and quality of life among elderly nursing home residents: Randomized controlled trial. Arch Gerontol Geriatr. 2017 May-Jun;70:92-98. doi: 10.1016/j.archger.2017.01.008. Epub 2017 Jan 16. PMID 28110207
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Sheikh, J.I. and Yesavage, J.A. (1986) Geriatric Depression Scale (GDS): Recent evidence and development of a shorter version. Clinical Gerontology, 5, 165-173
- [Background] La prise en charge des personnes âgées dépendantes ; rapport parlementaire présenté par Valérie Rosso-Debord ; Assemblée Nationale du 23 juin 2010
- [Background] Etat des lieux et préconisations sur l'hébergement temporaire des personnes âgées et des personnes handicapées ; CNSA ; Octobre 2011
- [Background] Évaluation des technologies de santé à la HAS : place de la qualité de vie ; Note de synthèse ; HAS
- [Background] Quelle qualité de vie ? Groupe OMS Qualité de Vie ; Forum mondial de la Santé, Volume 17, 1996
- [Background] Integrated Care for Older People: Guidelines on Community-Level Interventions to Manage Declines in Intrinsic Capacity. Geneva: World Health Organization; 2017. Available from http://www.ncbi.nlm.nih.gov/books/NBK488250/ PMID 29608259